

| Titolo | The role of <u>Surgery</u> in patients with CO <u>V</u> ID-19 related <u>Thor</u> acic <u>Co</u> mplications |
|---|---|
| Acronimo | SThor-CoV-2 |
| Versione del protocollo | V. 1.0 |
| Data del protocollo | 01/06/2021 |
| Tipologia di studio | Studio clinico osservazionale retrospettivo |
| Status del documento | Finale |
| Promotore | Università degli studi di Milano-Bicocca,<br>Dipartimento di Medicina e Chirurgia |
| Responsabile scientifico | Dr. Marco Scarci, UOC Chirurgia Toracica, ASST Monza, Ospedale San Gerardo, Monza, Italia, m.scarci@asst-monza.it |
| Project Manager | Dr. Federico Raveglia, UOC Chirurgia Toracica, ASST Monza, Ospedale San Gerardo, Monza, Italia, federico.raveglia@asstmonza.it |
| Amministratore del database | Dr. Arianna Rimessi, UOC Chirurgia Toracica, ASST Monza, Ospedale San Gerardo, Monza, Italia, <a href="mailto:arianna.rimessi@asst-monza.it">arianna.rimessi@asst-monza.it</a> Dr. Riccardo Orlandi, UOC Chirurgia Toracica, ASST Monza, Ospedale San Gerardo, Monza, Italia, riccardo.orlandi@unimi.it |
| Statistico | Prof. Paola Rebora, Statistica Medica, Università degli studi di Milano-Bicocca, Dipartimento di Medicina e Chirurgia, Monza, Italia, paola.rebora@unimib.it |

### Confidentiality statement:

Questo documento contiene informazioni riservate appartenenti all'Università di Milano-Bicocca. Ad eccezione di quanto diversamente concordato per iscritto, accettando o rivedendo questi materiali, l'utente accetta di conservare tali informazioni in modo confidenziale e di non rivelarle ad altri (salvo laddove richiesto dalla legge applicabile), né di usarli per scopi non autorizzati. In caso di effettiva o presunta violazione di tale obbligo, l'Università di Milano Bicocca deve essere tempestivamente informata.

## A D D O D I B I C O C A

### PROTOCOLLO DELLO STUDIO [SThor-CoV-2]

### - PAGINA DELLE FIRME

| Responsabile scientifico dello studio | |
|--------------------------------------------|------|
| Nome e Cognome: Marco Scarci | |
| Titolo accademico: Dottore | |
| Dipartimento: Cardio-Toraco-Vascolare | |
| Istituto: ASST Monza, Ospedale San Gerardo | |
| Città, Nazione: Monza, Italia | |
| Firma | Data |
| Principal investigator al centro | |
| Nome e Cognome: Federico Raveglia | |
| Titolo accademico: Dottore | |
| Dipartimento: Cardio-Toraco-Vascolare | |
| Istituto: ASST Monza, Ospedale San Gerardo | |
| Città, Nazione: Monza, Italia | |
| Firma | Data |

# BICOCCA

### PROTOCOLLO DELLO STUDIO [SThor-CoV-2]

### Sinossi

| Titolo dello studio | The role of <u>Surgery</u> in patients with CO <u>V</u> ID-19 related <u>Thor</u> acic <u>Co</u> mplications |
|---|---|
| Acronimo | SThor-CoV-2 |
| Background | Sempre più autori concordano sul fatto che gli interventi chirurgici elettivi debbano essere rinviati in caso di positività al SARS-CoV-2 a causa dell'incrementata morbi-mortalità peri-operatoria di questi pazienti. Sfortunatamente, vi è carenza di studi sull'efficacia e sulla sicurezza di un approccio chirurgico nella gestione di alcune possibili complicanze toraciche del COVID-19. In una recente pubblicazione tipo case-series, alcuni autorevoli ricercatori hanno descritto come fattibile la gestione chirurgica di alcune complicanze toraciche del COVID-19, registrando una sopravvivenza del 77%. |
| Razionale | Essendo il SARS-CoV-2 un virus prettamente respiratorio, le complicanze polmonari sono le più frequenti; alcune di queste potrebbero giovarsi di un trattamento chirurgico. Purtroppo, in letteratura, non esistono studi che forniscano indicazioni in questa direzione. Attraverso questo studio si cercherà di valutare se può avere senso operare pazienti con complicanze toraciche COVID-relate. |
| Obiettivo dello studio | Valutare l'efficacia e la sicurezza della gestione chirurgica delle complicanze toraciche COVID-relate |
| Disegno dello studio | Studio osservazionale retrospettivo multicentrico internazionale |
| Centri coinvolti | <ul> <li>Ospedale San Gerardo, Monza, Italia (centro coordinatore);</li> <li>Ospedale San Giovanni Battista Molinette, Torino, Italia;</li> <li>Ospedale Spedali Civili, Brescia, Italia;</li> <li>Ospedale San Camillo Forlanini, Roma, Italia;</li> <li>Ospedale University College London Hospitals, Londra, Regno Unito;</li> <li>Ospedale NYU Langone Health, New York, USA;</li> <li>Ospedale Hospital Federal do Andaraí, Rio de Janeiro, Brasile;</li> <li>Ospedale Chest Hospital, Calicut, India;</li> <li>Ospedale Sir Ganga Ram Hospital, New Delhi, India.</li> </ul> |
| Dimensione del campione | La dimensione campionaria attesa consta di circa 80 pazienti |
| Popolazione oggetto dello studio | Pazienti ricoverati con polmonite COVID-19 dal 01/03/2020 al 31/05/2021 che hanno sviluppato complicanze toraciche gestite mediante intervento chirurgico. |



| Principali criteri di | 1. Qualsiasi genere; |
|---|---|
| inclusione | 2. Età > o uguale a 18 anni; |
| | <ol> <li>Diagnosi virologica dell'infezione da SARS-CoV-2 attraverso<br/>real-time PCR;</li> </ol> |
| | Ricovero in ospedale a causa della diagnosi clinica/strumentale di polmonite; |
| | <ol> <li>Insorgenza di complicanza toracica durante il ricovero (nel<br/>caso di pazienti ospedalizzati) o che ha richiesto il ricovero<br/>(nel caso di pazienti al domicilio), per cui il paziente è stato<br/>sottoposto a intervento di chirurgia toracica;</li> </ol> |
| | 6. Periodo temporale dal 01/03/2020 al 31/05/2021. |
| Principali criteri di<br>esclusione | <ol> <li>Mancanza di diagnosi virologica di infezione da SARS-CoV-<br/>2 attraverso real-time PCR;</li> </ol> |
| | 2. Ricovero e intervento chirurgico oltre la <i>dead-line</i> 31/05/2021; |
| | 3. Pazienti con COVID-19 senza complicanze toraciche; |
| | <ol> <li>Complicanze toraciche che non hanno richiesto intervento<br/>chirurgico, ad esempio pneumotoraci gestiti<br/>conservativamente mediante l'esclusivo posizionamento di<br/>drenaggi pleurici.</li> </ol> |
| Endpoint primario | Sopravvivenza a 30 giorni dall'intervento. |
| p | Morbilità a 30 giorni dall'intervento. |
| Principali dati raccolti | Dati anagrafici; |
| | Dati anamnestici; |
| | Data diagnosi COVID-19; |
| | Complicanza necessitante intervento chirurgico; |
| | Data intervento chirurgico; |
| | Tipo di intervento chirurgico; |
| | Complicanze post-operatorie; |
| | Data di dimissione o exitus; |
| | Durata degenza; |
| | Causa di morte; |
| | Follow-up a 30 giorni (stato in vita e complicanze post-<br>operatorie) |

Acronimo:

# A D D C C C A ONE TIME IC O C C A

### PROTOCOLLO DELLO STUDIO [SThor-CoV-2]

| Metodi statistici | Misure di tendenza centrale e di dispersione saranno utilizzate per analisi descrittive. La sopravvivenza a 30 giorni sarà stimata con lo stimatore di Kaplan-Meier. Modelli di regressione logistica multipla saranno utilizzati allo scopo di identificare le variabili associate |
|---|---|
| | alla mortalità a 30 giorni dall'intervento e alle |
| | complicanze post-operatorie. |



### 1. INDICE

| Sinossi | 3 |
|------------------------------------------------------|----|
| 1. INDICE | 6 |
| 2. FLOWCHART | 7 |
| 3. BACKGROUND | 8 |
| 4. RAZIONALE | 8 |
| 5. OBIETTIVI ED ENDPOINTS | 9 |
| 6. CRITERI DI SELEZIONE DEI PAZIENTI | 9 |
| 6.1 Criteri di inclusione | 9 |
| 6.2 Criteri di esclusione | 9 |
| 7. DISEGNO DELLO STUDIO: | 10 |
| 7.1 Procedure studio specifiche | 10 |
| 7.2 Definizione di End of Study | 10 |
| 8. ANALISI STATISTICA | 11 |
| 9. PUBBLICAZIONE DEI RISULTATI | 11 |
| 10. ASPETTI ETICO/LEGALI | 11 |
| 10.1 Approvazione AC/CE | 11 |
| 10.2 Consenso informato | 11 |
| 10.3 Procedure di arruolamento | 12 |
| 10.4 Trattamento dei dati personali | 12 |
| 11. RACCOLTA, GESTIONE E CONSERVAZIONE DEI DATI: CRF | 12 |
| 11.1 Raccolta e gestione dei dati | 12 |
| 11.2 Conservazione dei dati | 14 |
| 12. CONTROLLO E ASSICURAZIONE DELLA QUALITA' | 14 |
| 13. BIBLIOGRAFIA | 15 |



### 2. FLOWCHART



<sup>\*</sup> Numero pazienti attesi, considerando arruolamento di circa 9 pazienti per centro.



### 3. BACKGROUND

COVID-19 è una patologia pandemica, che sta avendo un impatto devastante sulla vita di tutti i giorni e un peso senza precedenti sul nostro sistema sanitario [1]. Giorno dopo giorno, assistiamo ad un progressivo aumento di letteratura scientifica riguardante la patogenesi, le caratteristiche cliniche e i possibili trattamenti medici di questa patologia [2-5]. Con il passare del tempo, COVID-19 si è rivelata una patologia multisistemica, associata a complicanze che possono interessare pressocché ogni organo [6]. Questo ampio spettro di complicanze rende ragione dell'alto tasso di mortalità nei pazienti con comorbilità, il cui fragile equilibrio viene facilmente distorto dalla tempesta disimmune causata dal SARS-CoV-2 [7]. I pazienti "chirurgici" sono per loro natura fragili, a causa dell'importante stress esercitato dall'intervento chirurgico sull'omeostasi dell'organismo. Questo rende ragione degli outcomes peggiori rilevati nei pazienti con infezione da SARS-CoV-2 sottoposti ad interventi chirurgici in urgenza/emergenza [8, 9]. Diverse linee guida sono state pubblicate per cercare di regolamentare queste procedure chirurgiche, che per definizione non possono essere procrastinate. [10, 11]. In questo contesto, sempre più autori concordano sul fatto che gli interventi chirurgici elettivi debbano essere rinviati in caso di positività al SARS-CoV-2 a causa dell'incrementata morbi-mortalità perioperatoria di questi pazienti, soprattutto dal punto di vista respiratorio [12-18]. Tra le complicanze dell'infezione da SARS-CoV-2 potrebbero però essercene alcune meritevoli di un trattamento chirurgico. Sfortunatamente, vi è carenza di studi sull'efficacia e sulla sicurezza di un approccio chirurgico nella gestione di alcune possibili complicanze toraciche del COVID-19 come pneumotoraci, emotoraci, necrosi polmonare, empiemi, pneumatoceli e simili, limitandosi a singoli e isolati case report [19-23]. In una recente pubblicazione tipo case-series [24], alcuni autorevoli ricercatori hanno descritto come fattibile la gestione chirurgica di alcune complicanze toraciche del COVID-19, basandosi su una casistica di 13 pazienti e registrando una sopravvivenza del 77%. Partendo da questo presupposto, abbiamo organizzato uno studio multicentrico internazionale retrospettivo, analizzando tutti i pazienti affetti da COVID-19 che hanno sviluppato complicanze richiedenti un intervento di chirurgia toracica, nell'arco di tempo dal 01/03/2020 al 31/05/2021.

#### 4. RAZIONALE

Nei mesi trascorsi, ci siamo spesso scontrati con il problema dell'operabilità dei pazienti COVID-19, e verosimilmente ci troveremo sempre più a dover fronteggiare la questione con la progressiva endemizzazione del SARS-CoV-2. Essendo un virus prettamente respiratorio, le complicanze polmonari sono le più frequenti; alcune di queste potrebbero giovarsi di un trattamento chirurgico. Purtroppo, in letteratura, non esistono studi che forniscano indicazioni in questa direzione. Attraverso questo studio si cercherà di valutare se può avere senso operare pazienti con complicanze toraciche COVID-relate, indagando in via esplorativa quanti e quali fattori prognostici possano guidare la scelta di operare o meno il paziente

Acronimo:



### 5. OBIETTIVI ED ENDPOINTS

#### **OBIETTIVI**

#### Obiettivo primario

Valutare l'efficacia e la sicurezza della gestione chirurgica delle complicanze toraciche COVID-relate, confrontando gli outcomes di questi pazienti con quelli presenti in letteratura dei pazienti con analoghe complicanze, ma non COVID-relate, gestite chirurgicamente

#### Obiettivi secondari

Indagare i possibili fattori prognostici di questi pazienti sulla sopravvivenza a 30 giorni dall'intervento e sulle complicanze post-operatorie.

#### **ENDPOINTS**

#### **Endpoint primario**

Sopravvivenza a 30 giorni dall'intervento.

Morbilità a 30 giorni dall'intervento.

#### 6. CRITERI DI SELEZIONE DEI PAZIENTI

### 6.1 Criteri di inclusione

- Qualsiasi genere;
- 2. Età > o uguale a 18 anni;
- 3. Diagnosi virologica dell'infezione da SARS-CoV-2 attraverso real-time PCR;
- 4. Ricovero in ospedale a causa della diagnosi clinica/strumentale di polmonite;
- 5. Insorgenza di complicanza toracica durante il ricovero (nel caso di pazienti ospedalizzati) o che ha richiesto il ricovero (nel caso di pazienti al domicilio), per cui il paziente è stato sottoposto a intervento di chirurgia toracica;
- 6. Periodo temporale dal 01/03/2020 al 31/05/2021;

#### 6.2 Criteri di esclusione

- 1. Mancanza di diagnosi virologica di infezione da SARS-CoV-2 attraverso real-time PCR:
- 2. Ricovero e intervento chirurgico oltre la *dead-line* 31/05/2021;
- 3. Pazienti con COVID-19 senza complicanze toraciche;
- Complicanze toraciche che non hanno richiesto intervento chirurgico, ad esempio pneumotoraci gestiti conservativamente mediante l'esclusivo posizionamento di drenaggi pleurici;



#### 7. DISEGNO DELLO STUDIO:

Si tratta di uno studio clinico osservazionale retrospettivo multicentrico internazionale. I centri sono distribuiti in modo da coprire 5 differenti nazioni in 3 continenti, diversamente colpite dalla pandemia del SARS-CoV-2 e variabilmente organizzate per gestirla, così da poter avere dati scevri da influenze puramente territoriali, bensì generalizzabili su scala mondiale.

La popolazione oggetto di studio è costituita da tutti i pazienti ricoverati con polmonite COVID-19 dal 01/03/2020 al 31/05/2021 presso i centri partecipanti, che hanno sviluppato complicanze toraciche gestite mediante intervento chirurgico, che soddisfino tutti i criteri di inclusione, non presentando alcun criterio di esclusione.

Lo studio adotta un disegno longitudinale, con recupero retrospettivo dei dati relativi alle caratteristiche cliniche dei pazienti, alle complicanze legate al COVID-19 e agli interventi chirurgici eseguiti, e valutazione della sopravvivenza a 30 giorni dall'intervento e delle possibili complicanze post-operatorie.

### 7.1 Procedure studio specifiche

L'arruolamento dei pazienti avverrà retrospettivamente, selezionando i pazienti rispondenti ai criteri di inclusione nell'arco di tempo prestabilito. Per i pazienti risultati idonei, si procederà con la raccolta dei dati necessari e con la loro immissione in un database predisposto ad hoc. In considerazione della natura retrospettiva, lo studio non comporterà alcuna modifica della normale pratica clinica. Anche il follow-up a 30 giorni richiesto, consistente in una visita ambulatoriale con Rx torace di controllo, raccolta anamnestica ed esame obiettivo, rientrerà infatti nella normale prassi di rivalutazione postoperatoria dei pazienti sottoposti ad intervento chirurgico nei centri coinvolti nello studio.

### 7.2 Definizione di End of Study

Lo studio sarà concluso un mese dopo il termine della raccolta dati dei pazienti arruolati. Tale periodo si ritiene necessario per l'analisi dei dati raccolti.

### 8. ANALISI STATISTICA

Basandoci sul periodo di reclutamento e sui centri coinvolti ci attendiamo un campione di 80 soggetti. Questa numerosità campionaria ci permetterà di stimare la sopravvivenza a 30 giorni con una precisione di 0.194 (ampiezza totale dell'intervallo di confidenza con livello del 95%) assumendo una sopravvivenza di 0,770 [24]. Assumendo una possibile mancanza di dati per circa il 10% dei pazienti l'ampiezza totale dell'intervallo di confidenza con livello del 95% attesa sarebbe di 0.205 [25].

Misure di tendenza centrale e di dispersione saranno utilizzate per le analisi descrittive. La sopravvivenza a 30 giorni sarà stimata con lo stimatore di Kaplan-Meier. La sopravvivenza sarà stimata anche entro diagnosi e tipo di intervento chirurgico.



Modelli di regressione logistica multipla [26, 27] saranno utilizzati allo scopo di identificare le variabili associate alla mortalità a 30 giorni dall'intervento e alle complicanze post-operatorie. In particolare si valuteranno l'età, il fumo, la durata della degenza preoperatoria e il massimo supporto ventilatorio adottato.

#### 9. PUBBLICAZIONE DEI RISULTATI

Il responsabile scientifico dello studio si impegnerà nella stesura di un rapporto finale e di un articolo scientifico e a rendere pubblici i risultati al termine dello studio. I dati saranno resi pubblici in modo anonimo e presentati per quanto richiesto in modalità aggregata. La pubblicazione dei dati avverrà esclusivamente per fini scientifici, con l'intenzione di incrementare le conoscenze tecnico-teoriche del mondo scientifico sull'argomento, senza alcuno scopo di lucro.

#### 10. ASPETTI ETICO/LEGALI:

### 10.1 Approvazione AC/CE

Una copia del consenso informato del paziente deve essere sottomessa al CE insieme al protocollo per approvazione scritta. L'approvazione scritta del protocollo e del consenso informato devono essere ottenute prima di iniziare il reclutamento dei pazienti nello studio.

Il parere favorevole del Comitato Etico locale (CE) deve essere ottenuto prima dell'inizio della sperimentazione.

Il ricercatore deve informare il CE di eventuali emendamenti al protocollo, che devono essere approvati da quest'ultimo.

### 10.2 Consenso informato

Il PI prepara il consenso informato che verrà sottoposto al paziente appena se ne presenterà l'occasione. Qualora tale occasione non dovesse presentarsi non sarà necessario raccogliere il consenso informato del paziente in conformità all' articolo 89 del GDPR e all' Art. 11 comma 5 dell'allegato 1 (Codice di deontologia e di buona condotta per i trattamenti di dati personali per scopi statistici e scientifici) del provvedimento del Garante della privacy del 19/12/2018 n° 514 che recita: "il consenso dell'interessato non è necessario quando, sono soddisfatti i seguenti requisiti: a) non è possibile informare l'interessato per motivi etici (ignoranza dell'interessato sulla propria condizione), ovvero per motivi metodologici (necessità di non comunicare al soggetto le ipotesi dello studio o la sua posizione di elezione), ovvero per motivi di impossibilità organizzativa; b) il programma di ricerca è stato oggetto di motivato parere favorevole del competente comitato etico; c) il trattamento è autorizzato dal Garante, anche ai sensi dell'art. 40 del decreto anche su proposta di enti e società scientifiche pertinenti."

Acronimo:



#### 10.3 Procedure di arruolamento

Saranno arruolati tutti i soggetti che soddisfino i criteri di inclusione ed esclusione. In considerazione della natura retrospettiva osservazionale dello studio, i dati saranno raccolti e i pazienti selezionati retrospettivamente.

### 10.4 Trattamento dei dati personali

I dati personali oggetto dello studio dovranno essere trattati nel rispetto del Regolamento Europeo sulla Protezione dei Dati Personali (GDPR), del D.Lgs. 196/2003 e successive modifiche e integrazioni, e di ogni altra legge italiana applicabile alla protezione dei dati personali (da cui in poi definito come "legge per la protezione dei dati applicabile").

Relativamente ai dati personali resi disponibili al Promotore in forma pseudo anonimizzata, l'Istituto e il Promotore sono considerati cotitolari del trattamento dei dati, e entrambi agiranno in rispetto della legge per la protezione dei dati applicabile.

Inoltre, l'Istituto e il Promotore coopereranno per prendere le misure necessarie al fine di rispettare la legge per la protezione dei dati applicabile, e dovranno altresì implementare misure tecniche e organizzative appropriate per garantire i requisiti di conformità al GDPR.

L' Istituto è responsabile di fornire ai propri Principal Investigators e al Personale di ricerca tutte le informazioni necessarie relative alle modalità attraverso le quali il Promotore eventualmente raccoglierà e gestirà i loro dati personali prima che tali informazioni vengano fornite.

Il Promotore assicura la correttezza del trattamento dei dati personali come previsto dal GDPR. Se l'utente dovesse venire a conoscenza di un data breach di dati personali, l'utente stesso dovrà tempestivamente notificare agli altri utenti tale evento, e comunque entro e non oltre le 24 ore dall'avvenuta conoscenza dell'evento. In tal caso, l'utente dovrà cooperare pienamente con gli altri utenti per rimediare al data breach, adempiendo alla notifica obbligatoria nei tempi prestabiliti e gestendo l'eventuale danno causato.

Il data breach di dati personali è definito dagli art. 33 e 34 del GDPR.

### 11. RACCOLTA, GESTIONE E CONSERVAZIONE DEI DATI: CRF

#### 11.1 Raccolta e gestione dei dati

Lo studio verrà condotto nel rispetto dei dettami della dichiarazione di Helsinki e in accordo con le norme di una buona pratica clinica (D.M. Sanità del 15/07/1997 e s.m.i.) nonché con le disposizioni normative applicabili.

Ogni centro partecipante manterrà le cartelle cliniche e I dati di ricerca di questo studio in maniera appropriata, in conformità con la sezione 4.9 delle ICH-GCP E6, con le disposizioni degli enti regolatori e dell'istituzione di appartenenza per garantire la protezione della confidenzialità dei pazienti. In quanto partecipante ad uno studio clinico, ogni centro permetterà al personale autorizzato dallo sponsor e alle agenzie regolatorie di esaminare (e quando permesso dalla legge, di copiare) le cartelle cliniche allo scopo

Acronimo:



di controllare la qualità dei dati, per audit e per valutazioni della sicurezza e dello stato di avanzamento dello studio.

Documenti sorgente sono tutte le informazioni, record originali dei riscontri clinici, osservazioni, o altre attività di uno studio clinico necessarie alla ricostruzione e valutazione dello studio stesso. Esempi di questi documenti originali e record includono, ma non sono limitati a, cartelle cliniche, grafici clinici, quaderni di laboratorio, memoranda, diari dei pazienti o liste di valutazione, registri della dispensazione dei farmaci, dati registrati da strumenti automatici, copie o trascrizioni certificate dopo verifica che queste siano accurate e complete, microfiche, negativi fotografici, microfilm o supporti magnetici, lastre ottenute con raggi x, schede dei soggetti e registri tenuti nelle farmacie, nei laboratori, e nei dipartimenti tecnico-medici coinvolti nello studio clinico.

La raccolta dei dati è responsabilità del personale al centro coinvolto nello studio clinico sotto la supervisione del Principal Investigator del centro. La scheda di raccolta dati (CRF) è lo strumento principale per la raccolta dei dati dello studio. Il ricercatore dovrebbe garantire l'accuratezza, la completezza, la leggibilità e la tempestività dei dati riportati nella CRF e allo stesso modo degli altri dati riportati. I dati riportati nella CRF, che derivano da documenti sorgente, devono essere identici a quelli originali e dove così non fosse, la discrepanza dovrà essere spiegata. Tutti i dati richiesti dalla CRF dovranno essere registrati. Ogni dato mancante dovrà essere spiegato. Ogni cambiamento o correzione ad una CRF cartacea dovrà essere datata, riportate accanto le iniziali del compilatore, spiegata (se necessario) e non dovrà oscurare il dato originale. Il ricercatore dovrebbe tenere traccia dei cambiamenti e delle correzioni fatte alle CRF.

Il ricercatore/ istituzione dovrebbe mantenere I documenti dello studio come specificato in Documenti essenziali per la conduzione di uno studio clinico (ICH-GCP E6, sezione 8) e come richiesto dagli enti regolatori e/o dalle linee guida. Il ricercatore/ istituzione dovrebbe prendere misure per prevenire la distruzione accidentali o prematura della documentazione.

I documenti essenziali (scritti e elettronici) dovrebbero essere conservati per un periodo di tempo non inferiore a quindici (15) anni dal completamento dello studio, a meno che il Promotore fornisca un documento scritto che permetta di disporre e/o conservare i dati per un periodo di tempo aggiuntivo se permesso dalla legge, dagli enti regolatori e/o dalle linee quida.

I dati verranno raccolti mediante utilizzo di CRF cartacea.

I dati saranno raccolti in forma pseudo anonimizzata, ovvero per ogni soggetto verrà generato un codice alfa numerico (codice del soggetto) composto dal codice del centro, da un carattere spaziatore e dal numero del soggetto (es. CTR01-01) e i dati verranno archiviati elettronicamente.

Per tenere traccia dell'associazione tra cartella clinica e codice del soggetto, ogni centro compilerà un registro dove verranno riportati: codice del soggetto, nome e cognome, data di nascita e data dello screening. Tale registro, se in forma cartacea, dovrà essere conservato in un luogo ad accesso limitato e chiuso a chiave; se in forma elettronica, dovrà essere conservato in un file separato, criptato (crittografia AES-256) e protetto da

13/17

## DEGLI STUDIO DI BIO DI

### PROTOCOLLO DELLO STUDIO [SThor-CoV-2]

password; questo registro non verrà mai condiviso con il Promotore, né tanto meno con l'amministratore del database e nemmeno con lo statistico dello studio.

Nell'ambito dello studio verranno raccolti i seguenti dati:

- Informazioni anagrafiche
  - o Età
  - o Sesso
- Informazioni anamnestiche
  - Storia di fumo
  - o BPCO/asma
  - o Diabete mellito
  - o Insufficienza renale
  - Patologie cardiovascolari
  - Ipertensione polmonare
- Informazioni relative al ricovero per COVID-19
  - Data di diagnosi COVID-19
  - Utilizzo eparina
  - Ventilazione
  - o Posizionamento drenaggio pleurico
  - Imaging TC
  - Embolia polmonare
- Informazioni relative all'intervento chirurgico
  - o Giorno di intervento chirurgico
  - Diagnosi per l'intervento chirurgico
  - o Tipo di intervento chirurgico e tecnica adottata
  - Eventuali ulteriori interventi chirurgici
  - Ricovero in terapia intensiva
  - o Utilizzo ECMO
  - o Complicanze e rispettivo grado Clavien con intervento correttivo
  - Giorni di degenza post-operatori
  - o Causa e data di morte
  - Follow-up a 30 giorni (stato in vita e complicanze).

#### 11.2 Conservazione dei dati

La documentazione sarà disponibile, per eventuali controlli o ispezioni, per almeno 15 anni dalla chiusura formale dello studio. La conservazione dei dati avverrà a cura del responsabile scientifico.

### 12. CONTROLLO E ASSICURAZIONE DELLA QUALITA'

Presso ogni Centro verrà identificato un referente responsabile delle procedure di raccolta, verifica qualità e trasmissione dati. Le informazioni raccolte nei vari Centri Acronimo:



verranno periodicamente trasmesse al Centro Coordinatore (ASST Monza, Ospedale San Gerardo, Monza, Italia). Tali informazioni verranno inserite da personale addestrato in un database predisposto ad hoc dal Centro Coordinatore.

Ad ogni paziente verrà assegnato un codice unico identificativo, per garantirne l'anonimato. Lo sperimentatore del centro deve mantenere e custodire la corrispondenza tra le generalità del singolo pazienti inserito e il suo codice identificativo. Verranno registrati tutti gli eventi verificatisi durante il follow-up.

#### 13. BIBLIOGRAFIA

- 1. Shrestha N, Shad MY, Ulvi O, Khan MH, Karamehic-Muratovic A, Nguyen UDT, Baghbanzadeh M, Wardrup R, Aghamohammadi N, Cervantes D, Nahiduzzaman KM, Zaki RA, Haque U. The impact of COVID-19 on globalization. One Health. 2020 Dec 20;11:100180.
- 2. Yesudhas D, Srivastava A, Gromiha MM. COVID-19 outbreak: history, mechanism, transmission, structural studies and therapeutics. Infection. 2021 Apr;49(2):199-213.
- 3. Hu B, Guo H, Zhou P, Shi ZL. Characteristics of SARS-CoV-2 and COVID-19. Nat Rev Microbiol. 2021 Mar;19(3):141-154.
- 4. Salian VS, Wright JA, Vedell PT, Nair S, Li C, Kandimalla M, Tang X, Carmona Porquera EM, Kalari KR, Kandimalla KK. COVID-19 Transmission, Current Treatment, and Future Therapeutic Strategies. Mol Pharm. 2021 Mar 1;18(3):754-771.
- 5. Saito S, Asai Y, Matsunaga N, Hayakawa K, Terada M, Ohtsu H, Tsuzuki S, Ohmagari N. First and second COVID-19 waves in Japan: A comparison of disease severity and characteristics. J Infect. 2021 Apr;82(4):84-123.
- 6. Wiersinga WJ, Rhodes A, Cheng AC, Peacock SJ, Prescott HC. Pathophysiology, Transmission, Diagnosis, and Treatment of Coronavirus Disease 2019 (COVID-19): A Review. JAMA. 2020 Aug 25;324(8):782-793.
- 7. Chowdhury MA, Hossain N, Kashem MA, Shahid MA, Alam A. Immune response in COVID-19: A review. J Infect Public Health. 2020 Nov;13(11):1619-1629.
- 8. Colosimo C, Kelly J, Coker J, Bhuller S, Ballman E, Baker-Sparr C, Yon J, Cornett B, Dziadkowiec O, Weaver J. Unscreened: Urgent and Emergent Surgical Outcomes in the Early COVID-19 Pandemic. Cureus. 2020 Dec 3;12(12):e11878.
- 9. Knisely A, Zhou ZN, Wu J, Huang Y, Holcomb K, Melamed A, Advincula AP, Lalwani A, Khoury-Collado F, Tergas Al, St Clair CM, Hou JY, Hershman DL, D'Alton ME, Huang YY, Wright JD. Perioperative Morbidity and Mortality of



Patients With COVID-19 Who Undergo Urgent and Emergent Surgical Procedures. Ann Surg. 2021 Jan 1;273(1):34-40.

- 10. Coccolini F, Perrone G, Chiarugi M, Di Marzo F, Ansaloni L, Scandroglio I, Marini P, Zago M, De Paolis P, Forfori F, Agresta F, Puzziello A, D'Ugo D, Bignami E, Bellini V, Vitali P, Petrini F, Pifferi B, Corradi F, Tarasconi A, Pattonieri V, Bonati E, Tritapepe L, Agnoletti V, Corbella D, Sartelli M, Catena F. Surgery in COVID-19 patients: operational directives. World J Emerg Surg. 2020 Apr 7;15(1):25.
- 11. Coimbra R, Edwards S, Kurihara H, Bass GA, Balogh ZJ, Tilsed J, Faccincani R, Carlucci M, Martínez Casas I, Gaarder C, Tabuenca A, Coimbra BC, Marzi I. European Society of Trauma and Emergency Surgery (ESTES) recommendations for trauma and emergency surgery preparation during times of COVID-19 infection. Eur J Trauma Emerg Surg. 2020 Jun;46(3):505-510.
- 12.COVIDSurg Collaborative. Mortality and pulmonary complications in patients undergoing surgery with perioperative SARS-CoV-2 infection: an international cohort study. Lancet. 2020 Jul 4;396(10243):27-38.
- 13. De Luca M, Sartori A, Vitiello A, Piatto G, Noaro G, Olmi S, Foschi D, De Re L, Zappa M, Sarro G, Rivolta U, Giraudo G, Borghi F, Pozzo G, Sorisio V, Pignata G, Greco PA, Sisti V, Campagnaro T, Guglielmi A, Andreuccetti J, Di Leo A, Lauro E, Ricci F, Musella M, Zizzo M, Bonacini S, Podda M, Pisanu A, Coletta P, Guerrieri M, Caracino V, Basti M, Pilone V, Raffaelli M, Oragano L. Complications and mortality in a cohort of patients undergoing emergency and elective surgery with perioperative SARS-CoV-2 infection: an Italian multicenter study. Teachings of Phase 1 to be brought in Phase 2 pandemic. Updates Surg. 2021 Apr;73(2):745-752.
- 14. Kane AD, Paterson J, Pokhrel S, Berry SK, Monkhouse D, Brand JW, Ingram M, Danjoux GR. Peri-operative COVID-19 infection in urgent elective surgery during a pandemic surge period: a retrospective observational cohort study. Anaesthesia. 2020 Dec;75(12):1596-1604.
- 15. Prasad NK, Lake R, Englum BR, Turner DJ, Siddiqui T, Mayorga-Carlin M, Sorkin JD, Lal BK. Increased complications in patients who test COVID-19 positive after elective surgery and implications for pre and postoperative screening. Am J Surg. 2021 Apr 14:S0002-9610(21)00234-8.
- 16. Clement ND, Hall AJ, Makaram NS, Robinson PG, Patton RFL, Moran M, Macpherson GJ, Duckworth AD, Jenkins PJ. IMPACT-Restart: the influence of COVID-19 on postoperative mortality and risk factors associated with SARS-CoV-2 infection after orthopaedic and trauma surgery. Bone Joint J. 2020 Dec;102-B(12):1774-1781. doi: 10.1302/0301-620X.102B12.BJJ-2020-1395.R2. Epub 2020 Oct 21. PMID: 33249904.

Acronimo:



- 17. Salmerón Jiménez M, Hermoso Alarza F, Martínez Serna I, Marrón Fernández C, Meneses Pardo JC, García Salcedo JA, Torres Serna A, Manama Gama MG, Colmenares Mendoza OE, Diaz-Hellín Gude V, Gamez García AP. Clinical features and outcomes of thoracic surgery patients during the COVID-19 pandemic. Eur J Cardiothorac Surg. 2020 Oct 1;58(4):738-744.
- 18. Patriti A, Baiocchi GL, Catena F, Marini P, Catarci M; FACS on behalf of the Associazione Chirurghi Ospedalieri Italiani (ACOI). Emergency general surgery in Italy during the COVID-19 outbreak: first survey from the real life. World J Emerg Surg. 2020 May 24;15(1):36.
- 19. Aiolfi A, Biraghi T, Montisci A, Bonitta G, Micheletto G, Donatelli F, Cirri S, Bona D. Management of Persistent Pneumothorax With Thoracoscopy and Bleb Resection in COVID-19 Patients. Ann Thorac Surg. 2020 Nov;110(5):e413-e415.
- 20.Bellini R, Salandini MC, Cuttin S, Mauro S, Scarpazza P, Cotsoglou C. Spontaneous pneumothorax as unusual presenting symptom of COVID-19 pneumonia: surgical management and pathological findings. J Cardiothorac Surg. 2020 Oct 12;15(1):310.
- 21. Geraci T.C., Narula N., Smith D.E., Moreira A.L., Kon Z.N., Chang S.H. Lobectomy for hemorrhagic lobar infarction in a patient with COVID-19. Ann Thorac Surg. 2020;111:e183–e184.
- 22. Castiglioni M., Pelosi G., Meroni A., Tagliabue M., Uslenghi E., Salaris D. Surgical resections of superinfected pneumatoceles in a COVID-19 patient. Ann Thorac Surg. 2020;111:e23–e25.
- 23. Tessitore A, Patella M, Giuliani M, Theologou T, Freguia S, Minerva EM, Rugel G, Cafarotti S. Surgical treatment of pleural empyema in Coronavirus disease 19 patients: the Southern Switzerland experience. Interact Cardiovasc Thorac Surg. 2021 Apr 8;32(3):367-370.
- 24. Chang SH, Chen D, Paone D, Geraci TC, Scheinerman J, Bizekis C, Zervos M, Cerfolio RJ. Thoracic surgery outcomes for patients with Coronavirus Disease 2019. J Thorac Cardiovasc Surg. 2021 Jan 30:S0022-5223(21)00168-9.
- 25. Fleiss J.L., Levin B., Paik M.C. 2003. Statistical Methods for Rates and Proportions. Third Edition. John Wiley & Sons. New York.
- 26. McCullagh, P. Regression Models for Ordinal Data. Journal of the Royal Statistical Society. Series B (Methodological) 1980; 42(2):109-142.
- 27. Cox DR. Journal of the Royal Statistical Society. Series B (Methodological) 1972; 34(2):187- 220.